CLINICAL TRIAL: NCT05917093
Title: Culturally Tailoring the Delivery of an Evidence-Based Diabetes Self-Management Program for Black Adults to Enhance Its Reach, Adoption, Implementation, and Effectiveness
Brief Title: Healthy Living for You
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: UW Institute of Clinical and Translational Research (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-0821; Protocol Version 7/9/2024 (Other: UW Madison); PHARM/PHARMACY (Other: UW Madison)
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Diabetes
Keywords: diabetes self-management; cultural tailoring; Healthy Living with Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Culturally tailored HLWD (Experimental)
  Interventions: Behavioral: Culturally tailored HLWD

INTERVENTIONS:
Behavioral: Culturally tailored HLWD — Participants receive the culturally tailored HLWD intervention for 6 weeks
  * Week 0 - Baseline enrollment.
  * Weeks 1-6 will consist of 6 separate group sessions. Diabetes self-management topics will be covered by 2 Black HLWD Facilitators. Participants will meet once a week, for a 2½-hour session, in community settings such as a community center, or church.
  Other Names: Healthy Living With Diabetes

SUMMARY:
The goal of the study is to conduct the Healthy Living with Diabetes (HLWD) program among Black individuals in a culturally appropriate manner. This study will involve 24-30 participants in total. Participants can expect to be on study for approximately 6 months.

DETAILED DESCRIPTION:
The study objectives are to recruit and empower Black Healthy Living with Diabetes (HLWD) facilitators to deliver culturally tailored HLWD content and pilot the culturally tailored HLWD program, using the RE-AIM framework and Proctor implementation outcomes to gather preliminary implementation data. The study team will partner with stakeholders and community organizations serving Black adults, including Grace Fellowship Church and YMCA of Metropolitan Milwaukee. The central hypothesis is that the cultural tailoring of HLWD will increase the reach, adoption, implementation, and effectiveness of HLWD among Black adults.

The study aims are:

1. Co-design a culturally relevant approach to the recruitment and training of Black HLWD facilitators. The study team will partner with a stakeholder advisory board including:

   * (1) Black adults with diabetes (prior HLWD participants)
   * (2) Black community leaders
   * (3) current Black HLWD facilitators, and
   * (4) current HLWD program providers (organizational leaders in settings delivering HLWD to Black adults)

   to co-design: (a) an asset-based approach to recruiting Black facilitators and (b) an adjunct training that empowers the facilitator to use a culturally relevant approach to deliver HLWD content to Black adults.
2. Implement the culturally tailored HLWD program among Black adults. Using a mixed methods design, the investigators will assess recruitment/retention rates among Black adults (reach), feasibility of adoption among facilitators and program providers (adoption), participant adherence, fidelity of enactment and acceptability, fidelity of program delivery by facilitators (implementation), and pre-post impact on diabetes outcomes (effectiveness).

ELIGIBILITY:
Inclusion Criteria:

* self-identify as Black/African American
* have type 1 diabetes, type 2 diabetes, gestational diabetes, or pre-diabetes

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Recruitment: Number of HLWD Participants Enrolled in a HLWD Workshop vs Invited to Enroll | up to 6 months
Recruitment: Number of Miles Participants are Willing to Travel for a Workshop | up to 6 months
Summary of Reasons for Agreeing to Participate Reported by Participant Count | up to 6 months
  Qualitative measure where reasons will be coded and grouped into themes for reporting.
Summary of Reasons for Declining to Participate Reported by Participant Count | up to 6 months
  Qualitative measure where reasons will be coded and grouped into themes for reporting.
Retention: Proportion of Participants who Completed the HLWD Workshop and Final Assessments | up to 6 months
Retention Rate during a 6-week Session | Up to 6 weeks
Summary of Reasons for Dropping Out by Participant Count | up to 6 months
  Qualitative measure where reasons will be coded and grouped into themes for reporting.

SECONDARY OUTCOMES:
Effectiveness: Diabetes Empowerment Scale - Short Form Self-Efficacy for Adherence to Medication Use Scale | Baseline, 6 weeks, 6 months
  The Diabetes Empowerment Scale is a 8-item survey each scored on a 5 point likert scale. This scale assesses the patients' perceived ability to obtain social support, manage stress, be self-motivating and make diabetes-related decisions. A total range of score is from 0-40. Higher score indicate higher diabetes empowerment.
Effectiveness: Patient's Perceived Involvement in Care Scale (PICS) | Baseline, 6 weeks, 6 months
  PICS is a 13-item survey where each item is scored yes (1) or no (0) for a total range of scores from 0-13. This instrument is designed to examine three relatively distinct factors: (1) doctor facilitation of patient involvement, (2) level of information exchange, and (3) patient participation in decision making. Higher score indicate higher patient/provider communication quality.
Effectiveness: Self-Reported Health Status | Baseline, 6 weeks, 6 months
  Participants self-reported their overall health on a scale of by selecting one of the 5 options: poor, fair, good , very good, or excellent. Scoring is from 1-5 with higher scores indicating poor health.
Facilitator Adoption: Number Agreeing to be a Facilitator divided by the Number Approached | up to 6 months
Facilitator Evaluation Reported in binary Yes / No | up to 6 months
  Facilitators will be asked if they satisfied with the training and experience of being a facilitator? Would they consider leading another program? Would they recommend being a facilitator?
Facilitator Feedback | up to 6 months
  Qualitative measure to be coded and themed, summarizing barriers to adoption.
Implementation: Weekly Session Attendance | up to 6 weeks
Implementation: Summary of Diabetes Self-Care Activities (SDSCA) | up to 6 weeks
  The SDSCA is a 7-item survey with each item scored from 0-7. The total possible range of scores is from 0-112, with higher scores indicating better self-care.
Implementation: Participant Satisfaction Ratings | up to 6 weeks
  Participant Satisfaction Ratings are scored from 1-5, with higher scores indicating higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Chui, PharmD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - YMCA, Milwaukee, Wisconsin
  - Grace Fellowship Church, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/93/NCT05917093/ICF_000.pdf